CLINICAL TRIAL: NCT06808867
Title: A 6-week Randomized, Double-blind, Comparative Clinical Study of the Efficacy of an Oral Product in Subjects With Acid Reflux and/or Abdominal Bloating/Distention and Gastrointestinal Symptoms
Brief Title: Efficacy of Dietary Supplement in Subjects With Acid Reflux and/or Abdominal Bloating/Distention and GI Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olly, PBC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: UNLV20231116
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Oral dietary supplement. Instructions: Subjects were instructed to take the product (1 pill) with a glass of water in the morning.
  Interventions: Dietary Supplement: Placebo
- Dietary Supplement with Active Ingredient Blend (Active Comparator): Oral dietary supplement. Instructions: Subjects were instructed to take the product (1 pill) with a glass of water in the morning.
  Interventions: Dietary Supplement: Dietary Supplement with Active Ingredient Blend

INTERVENTIONS:
Dietary Supplement: Placebo — Eligible subjects will receive Placebo to take daily for six weeks
  Arms: Placebo
Dietary Supplement: Dietary Supplement with Active Ingredient Blend — Eligible subjects will receive Active supplement to take daily for six weeks
  Arms: Dietary Supplement with Active Ingredient Blend

SUMMARY:
This study was a prospective randomized clinical study. There was interventional treatment for a total of 8 weeks including a 2-week washout period. The subjects attended four appointments in the clinic throughout the duration of the study.

Study Primary Objective:

• To assess improvement in bloating symptoms

Study Secondary Objectives:

* To assess safety and tolerability of the formulation
* To compare the time taken for perceptual improvement in bloating/distention
* Enzyme blood assays
* To assess quality of life indices

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in the study.
* Willingness to actively participate in the study and to come to the scheduled visits.
* Female and/or male
* From 18 to 85 years of age
* Patients with self-reported abdominal bloating, abdominal distention, flatulence, and abdominal discomfort either after meals or not at least 3x a week for a minimum of the past 2 weeks

Exclusion Criteria:

* Drug addicts, alcoholics.
* AIDS, HIV-positive or infectious hepatitis
* Diabetes mellitus
* Disorders known to affect GI motility such as gastroparesis or amyloidosis.
* Disorders with GI symptoms such as irritable bowel syndrome, inflammatory bowel disease and celiac disease
* History of surgery known to alter the normal function of the GI tract.
* Conditions which exclude participation or might influence the test reaction/evaluation.
* Participation or being in the waiting period after participation in cosmetic and/or pharmaceutical studies pertaining to the test area.
* Cancer not being diagnosed as cured and requiring chemotherapy, irradiation and/or hormonal treatment within the last 2 years.
* Documented allergies to cosmetic products and/or ingredients
* Systemic therapy with immuno-suppressive drugs (e.g. corticosteroids) within the last 6 weeks prior to the start of the study and/or throughout the entire course of the study.
* Oral steroids within the last 4 weeks prior to the start of the study and/or throughout the entire course of the study
* Oral or systemic therapy with antibiotics within the last 3 months prior to the start of the study and/or throughout the entire course of the study
* Subjects who were treated with biologics within the last 6 months prior to the start of the study and/or throughout the entire course of the study.
* One of the following illnesses if not medicated: cardiovascular diseases, thyroid hyperfunction, asthma, hypertension.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2024-02-25 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Changes in Digestive Quality of Life Questionnaire (DQLQ) scores | from enrollment to end of study at 8 weeks
  To assess changes in scores related to bloating, diarrhea, constipation and heartburn on quality-of-life indicators, comparing active supplement to placebo group
Changes in Symptom Severity Score (Diary) | from enrollment to end of study at 8 weeks
  Patients filled out the symptoms diary that had questionnaires of bowel habits. Abdominal pain and bloating were rated on a 100-point visual analogue scale with 0=none and 100=severe, comparing active supplement to placebo group

SECONDARY OUTCOMES:
Changes in Gastrointestinal Short Form Questionnaire (GSFQ) Scores | from enrollment to end of study at 8 weeks
  To assess changes in gastrointestinal symptoms comparing active supplement to placebo group
Changes in Stool Consistency (Bristol Stool Scale) | from enrollment to end of study at 8 weeks
  Daily stool consistency ratings will provide data on changes in bowel health and regularity. Average stool consistency scores will be compared across baseline, active treatment, and placebo phases.

CONTACTS AND LOCATIONS:
Locations (1):
- See Final Report, San Francisco, California, United States